CLINICAL TRIAL: NCT00130780
Title: Multimodality Treatment for Patients With Resectable Non-Small Cell Lung Cancer (NSCLC) (BEACON Study: Bevacizumab and Chemotherapy for Operable NSCLC)
Brief Title: Multimodality Treatment for Patients With Resectable Non-Small Cell Lung Cancer (NSCLC) - BEACON Study: Bevacizumab and Chemotherapy for Operable NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-052
Record Dates: First submitted 2005-08-12; First posted 2005-08-16 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Multi-modality treatment for lung cancer; Carcinoma, Squamous Cell; Bevacizumab; BEACON; 05-052
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell | interventions — Bevacizumab; Drug Therapy; Cisplatin

ARMS (2):
- A (Active Comparator): Pre-surgical Treatment with Bevacizumab plus Chemotherapy
  Interventions: Drug: Pre-surgical Treatment with Bevacizumab plus Chemotherapy
- B (Active Comparator): Pre-Surgical Docetaxel and Cisplatin and Adjuvant Bevacizumab
  Interventions: Drug: Pre-Surgical Docetaxel and Cisplatin and Adjuvant Bevacizumab

INTERVENTIONS:
Drug: Pre-surgical Treatment with Bevacizumab plus Chemotherapy — On Cycle 1 Day 1,patient will receive bevacizumab 15 mg/kg. On Cycle 1 Day 15, patients receive docetaxel (75 mg/m2), cisplatin (75 mg/m2). Cycle 2 begins 21 days after administration of docetaxel and cisplatin in Cycle 1. In Cycles 2 thru 3, patients will receive 2 preoperative 21-day cycles of docetaxel (75 mg/m2), cisplatin (75 mg/m2), and bevacizumab (15 mg/kg), all given on Day 1 of each cycle. The sequence of administration will be docetaxel, followed by cisplatin, followed by bevacizumab according to MSKCC Chemotherapy Guidelines. In Cycle 4 Day 1, patients will receive docetaxel (75 mg/m2) and cisplatin (75 mg/m2). Bevacizumab will not be given with Cycle 4. During Cycle 4, the only scheduled clinic visit will be on Day 1. Surgery will occur at least 42 days after the last treatment with bevacizumab. Every attempt will be made to administer the treatment on schedule. The treatment may be given +/- 3 days, and additionally 2 weeks after it is scheduled, if necessary.
  Arms: A
Drug: Pre-Surgical Docetaxel and Cisplatin and Adjuvant Bevacizumab — Patients will receive preoperative 21-day cycles of cisplatin (75 mg/m2) and docetaxel (75 mg/m2) both given on Day 1 of each cycle.Patients will undergo repeat CT imaging after 2 cycles of therapy and patients with at least 10% reduction in bidimensional tumor volume will receive 2 additional neoadjuvant cycles of therapy (total 4 cycles of therapy).Surgery will occur at least 4 weeks after the last treatment with docetaxel and cisplatin.Adjuvant bevacizumab (15 mg/kg q21 days for 1 year, total 18 cycles) will be administered to all patients who undergo resection. Adjuvant bevacizumab will begin between days 42 and 56 after surgery.Patients may be referred for post-operative radiation therapy at the discretion of the treating physician. Every attempt will be made to administer the treatment on schedule. The treatment may be given +/- 3 days, and additionally 2 weeks after it is scheduled, if necessary.
  Arms: B

SUMMARY:
This is a phase II, single institution trial for patients with clinical Stage IB-IIIA NSCLC (T1-3N0-2M0) who have resectable lung tumors. The primary goal of this study is to show that the addition of bevacizumab to a cisplatin-based chemotherapy in the neoadjuvant setting for non-squamous cell carcinomas improves the rate of pathologic downstaging, which correlates with survival. Downstaging is defined as any decrease in the final pathologic stage compared with the clinical stage before induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of NSCLC at Memorial Sloan-Kettering Cancer Center (MSKCC)
* Stages IB, IIA, IIB or IIIA (T1-3N0-2M 0) NSCLC
* Patients must be candidates for resection with curative intent.
* Measurable disease, defined as at least one lesion that can be accurately measured in at least two dimensions
* Age >= 18 years
* Karnofsky performance status >= 70%
* Normal marrow function: leukocytes >= 3,000/µl; absolute neutrophil count ≥ 1,500µl; platelets >= 100,000 µl; hemoglobin >= 9gm/dl.
* Adequate renal function, with creatinine <= 1.3 mg/dl or calculated creatinine clearance >= 60ml/min by Cockcroft-Gault equation using parameters of age, weight (kg), and baseline serum creatinine (mg/dl)
* Adequate hepatic function: total bilirubin within normal limits; AST <= 1.5 X upper limit of normal (UNL); ALT <= 1.5 X UNL; alkaline phosphatase <= 1.5 X UNL.
* Women of childbearing age must have a negative urine or blood pregnancy test.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Patients must have ability to understand and the willingness to sign a written informed consent document.
* Eligibility criteria for group B: Patients with SQUAMOUS CELL carcinoma or patients with a NON-SQUAMOUS CELL tumor with a large central tumor in proximity to significant blood vessels or any history of hemoptysis will be assigned to group B (preoperative chemotherapy alone without bevacizumab).

Exclusion Criteria:

* Prior chemotherapy or radiation therapy for NSCLC
* Prior treatment with bevacizumab or other agents specifically targeting vascular endothelial growth factor (VEGF)
* Patients with a history of severe hypersensitivity reaction to docetaxel (Taxotere) or other drugs formulated with polysorbate 80
* Patients with known hypersensitivity to other recombinant human antibodies
* Patients must not be receiving any other investigational agents.
* History of stroke or transient ischemic attack (TIA).
* History of myocardial infarction or unstable angina within the past 12 months.
* Patients who report a hearing deficit at baseline, even if it does not require a hearing aid or intervention, or interfere with activities of daily life (Common Terminology Criteria for Adverse Events [CTCAE] grade 2 or higher)
* Peripheral neuropathy > grade 1.
* Uncontrolled hypertension
* Esophageal varices, non-healing ulcer, wound, or bone fracture
* Known HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with the study drugs.
* Other serious illness or medical condition including unstable cardiac disease requiring treatment, history of significant neurologic or psychiatric disorders (including psychotic disorders, dementia, or seizures), symptomatic diverticulitis, or active uncontrolled infection.
* Women who are pregnant or breast-feeding
* Psychiatric illness or social situation that would limit compliance with study requirements
* Exclusion criteria for group A: Patients with SQUAMOUS CELL carcinoma, large central tumor in proximity to significant blood vessels, or any history of hemoptysis (will be excluded from group A (preoperative chemotherapy plus bevacizumab); these patients will be assigned to group B (preoperative chemotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2005-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naiyer Rizvi, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- A: Pre-surgical Treatment With Bevacizumab Plus Chemotherapy: Pre-surgical Treatment with Bevacizumab plus Chemotherapy
  Pre-surgical Treatment with Bevacizumab + Chemotherapy: On Cycle 1 Day 1,patient will receive bevacizumab 15 mg/kg. On Cycle 1 Day 15, patients receive docetaxel (75 mg/m2), cisplatin (75 mg/m2). Cycle 2 begins 21 days after administration of docetaxel and cisplatin in Cycle 1. In Cycles 2 thru 3, patients will receive 2 preoperative 21-day cycles of docetaxel (75 mg/m2), cisplatin (75 mg/m2), and bevacizumab (15 mg/kg), all given on Day 1 of each cycle. The sequence of administration will be docetaxel, followed by cisplatin, followed by bevacizumab according to MSKCC Chemotherapy Guidelines. In Cycle 4 Day 1, patients will receive docetaxel (75 mg/m2) and cisplatin (75 mg/m2). Bevacizumab will not be given with Cycle 4. During Cycle 4, the only scheduled clinic visit will be on Day 1. Surgery will occur at least 42 days after the last treatment with bevacizumab. Every attempt will be made to administer the treatment on sc
- B: Pre-Surgical Docetaxel, Cisplatin, and Adjuvant Bevacizumab: Pre-Surgical Docetaxel and Cisplatin and Adjuvant Bevacizumab
  Pre-Surgical Docetaxel and Cisplatin and Adjuvant Bevacizumab: Patients will receive preoperative 21-day cycles of cisplatin (75 mg/m2) and docetaxel (75 mg/m2) both given on Day 1 of each cycle.Patients will undergo repeat CT imaging after 2 cycles of therapy and patients with at least 10% reduction in bidimensional tumor volume will receive 2 additional neoadjuvant cycles of therapy (total 4 cycles of therapy).Surgery will occur at least 4 weeks after the last treatment with docetaxel and cisplatin.Adjuvant bevacizumab (15 mg/kg q21 days for 1 year, total 18 cycles) will be administered to all patients who undergo resection. Adjuvant bevacizumab will begin between days 42 and 56 after surgery.Patients may be referred for post-operative radiation therapy at the discretion of the treating physician. Every attempt will be made to administer the treatment on schedule. The treatment may be given +/- 3 days, and additionally
Period: Overall Study
Arm/Group | A: Pre-surgical Treatment With Bevacizumab Plus Chemotherapy | B: Pre-Surgical Docetaxel, Cisplatin, and Adjuvant Bevacizumab
Started | 51 | 20
Completed | 51 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Pre-surgical Treatment With Bevacizumab Plus Chemotherapy | B: Pre-Surgical Docetaxel, Cisplatin, and Adjuvant Bevacizumab | Total
Number analyzed (Participants) | 51 | 20 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 16 | 52
  >=65 years | 15 | 4 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 7 | 38
  Male | 20 | 13 | 33
Region of Enrollment [Number; unit: participants]
  United States | 51 | 20 | 71

OUTCOME MEASURES:

1. Primary Outcome: The Primary Goal of This Study is to Show That the Addition of Bevacizumab to Cisplatin-based Chemotherapy in the Neoadjuvant Setting for Non-squamous Cell Carcinomas Improves Therapeutic Response/Outcome Assessment.
Description: These criteria have been modified for the purpose of this study (i.e.: there will be no confirmation of response at 4 weeks per usual response criteria as this is not applicable to the preoperative treatment plan): Complete Response (CR): Disappearance of all clinical evidence of tumor. Partial Response (PR): A 50% or greater decrease in the sum of the products of measured lesions. No simultaneous increase in the size of any lesion or the appearance of new lesions may occur. Non-measurable lesions must remain stable or regress for this category. Minor Response (MR): A > 25% and < 50% decrease in the sum of the products of measured lesions. No simultaneous increase in the size of any lesion or the appearance of new lesions may occur. Non-measurable lesions must remain stable or regress for this category. Stable Disease (SD): A less than 25% decrease. This includes a decrease of less than 25% in the sum of the products of the meas
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | A: Pre-surgical Treatment With Bevacizumab Plus Chemotherapy | B: Pre-Surgical Docetaxel, Cisplatin, and Adjuvant Bevacizumab
Number analyzed (Participants) | 51 | 20
participants | 51 | 20

ADVERSE EVENTS:
Arm/Group | A: Pre-surgical Treatment With Bevacizumab Plus Chemotherapy | B: Pre-Surgical Docetaxel, Cisplatin, and Adjuvant Bevacizumab
Serious Adverse Events (participants affected / at risk) | 28/51 | 6/20
Other Adverse Events (participants affected / at risk) | 49/51 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Pre-surgical Treatment With Bevacizumab Plus Chemotherapy (N=51) | B: Pre-Surgical Docetaxel, Cisplatin, and Adjuvant Bevacizumab (N=20)
Dehydration (Gastrointestinal disorders) | 4 (5) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0)
Enteritis (inflamm of small bowel) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Mucositis (Clin exam)- Oral cavity (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 4 (4) | 2 (2)
Pain - Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Pre-surgical Treatment With Bevacizumab Plus Chemotherapy (N=51) | B: Pre-Surgical Docetaxel, Cisplatin, and Adjuvant Bevacizumab (N=20)
ALT, SGPT (Metabolism and nutrition disorders) | 1 (6) | 3 (10)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 18 (54) | 3 (8)
Bilirubin (hyperbilirubinemia) (Investigations) | 3 (17) | 1 (2)
Constipation (Gastrointestinal disorders) | 9 (13) | 1 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (11) | 2 (4)
Creatinine (Investigations) | 4 (10) | 2 (2)
Dehydration (Gastrointestinal disorders) | 2 (4) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (14) | 3 (6)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 1 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 34 (106) | 9 (20)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 40 (90) | 15 (41)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 13 (18) | 3 (6)
Hemoglobin (Blood and lymphatic system disorders) | 35 (79) | 11 (22)
Hypertension (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 15 (23) | 4 (6)
Lymphopenia (Investigations) | 15 (21) | 7 (14)
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 8 (12) | 2 (3)
Mucositis (Clin exam)- Oral cavity (Gastrointestinal disorders) | 12 (29) | 4 (5)
Nausea (Gastrointestinal disorders) | 13 (32) | 2 (6)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 20 (26) | 4 (4)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 13 (14) | 6 (6)
Platelets (Investigations) | 5 (8) | 0 (0)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 7 (10) | 0 (0)
Potassium, low (hypokalemia) (Investigations) | 3 (3) | 0 (0)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 9 (12) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 12 (19) | 4 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes